CLINICAL TRIAL: NCT04943159
Title: A Phase II, Randomised, Open Label Pilot Study to Evaluate the Efficacy and Safety of Two Dosage Regimens of Subcutaneous Bioresorbable Afamelanotide Implants in Patients With Mild to Moderate Acne Vulgaris
Brief Title: Afamelanotide in Patients Suffering With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUV100
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — afamelanotide

ARMS (2):
- Afamelanotide group A (Experimental)
  Interventions: Drug: Afamelanotide
- Afamelanotide group B (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide — Group A is administered afamelanotide implant on Days 0, 21 and 42; Group B is administered afamelanotide implant on Days 0 and 28.

SUMMARY:
This study aims to evaluate the effect of afamelanotide on the facial inflammatory acne-related lesions in patients with mild to moderate acne vulgaris, including tolerability of afamelanotide by patients with moderate acne vulgaris and effects of the treatment on quality of life in eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with a diagnosis of mild to moderate acne vulgaris, defined as an Investigator's global assessment (IGA) score of 2-3;
* Chronic course of acne vulgaris;
* Acne-related lesions both on the face, chest and back;
* Indication for treatment of acne vulgaris;
* Aged 18-30 years (inclusive);
* Fitzpatrick skin types I-III;
* Providing written Informed Consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* Female subjects;
* Diagnosis of severe acne vulgaris;
* Allergy to afamelanotide or the polymer contained in the implant or to lidocaine or other local anesthetic to be used during the administration of the implant;
* Use of topical acne medication such as retinoids, benzoyl peroxide or topical antibiotics within 2 weeks prior to the first dose;
* Use of oral antibiotics for acne within 4 weeks prior to the first dose;
* Use of topical corticosteroids on the face, chest and back or systemic corticosteroids within the past 4 weeks prior to the first dose;
* Use of systemic retinoids within 6 months prior to the first dose;
* Use of anti-androgenic agents such as finasteride within 4 weeks prior to the first dose;
* Use of phototherapy devices for acne such as ClearLight™ or Zenozapper within 1 week prior to the first dose;
* Use of tanning booths or lamps within 1 week prior to the first dose;
* Active skin disease that may interfere with evaluation;
* Other forms of acne such as acne rosacea, acne excoriée, chloracne, acne conglobata, acne fulminans, acne inversa or drug-induced acne;
* Participation in a clinical trial for an investigational agent within 30 days prior to the screening visit.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-08-24 (Actual); Primary Completion 2011-03-08 (Actual); Study Completion 2011-03-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A pooled analysis of all the patients treated by afamelanotide (group A and group B) was conducted as only 3 patients were recruited in the study (2 in group A and one in group B) due to difficulties in recruitment.
Groups:
- Afamelanotide (Pooled Analysis): * Group A are administered afamelanotide implant on Days 0, 21 and 42;
  * Group B are administered afamelanotide implant on Days 0 and 28.
Period: Overall Study
Arm/Group | Afamelanotide (Pooled Analysis)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A pooled analysis of all the patients treated by afamelanotide (group A and group B) was conducted as only 3 patients were recruited in the study (2 in group A and one in group B) due to difficulties in recruitment.
Arm/Group | Afamelanotide (Pooled Analysis)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: The Change in Number of Facial Inflammatory Acne-related Lesions.
Time Frame: From baseline to Day 56.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Lesions
Arm/Group | Afamelanotide (Pooled Analysis)
Number analyzed (Participants) | 3
Lesions
  Baseline | 46 (30.3)
  Day 56 | 23.7 (15.6)

ADVERSE EVENTS:
Description: A pooled analysis of all the patients treated by afamelanotide (group A and group B) was conducted as only 3 patients were recruited in the study (2 in group A and one in group B) due to difficulties in recruitment.
Arm/Group | Afamelanotide (Pooled Analysis)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (Pooled Analysis) (N=3)
Fatigue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No